CLINICAL TRIAL: NCT05874791
Title: Executive Control Training for Adolescents With ADHD: A Randomized Controlled
Brief Title: Executive Control Training for Adolescents With ADHD: A Randomized Controlled Effectiveness Trial
Acronym: ADHD Effect
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sykehuset Innlandet HF (Other)
Collaborators: University of Oslo (Other); Lovisenberg Diakonale Hospital (Other); Oslo University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 150687 and 150688; 420217 (Other: REK); 150688 (Other: Innlandet Hospital Trust (PhD)); 150687 (Other: Innlandet Hospital Trust (Post doc)); 102610213 (Other: Department of Psychology, University of Oslo (PhD)); 103876101 (Other: Oslo University Hospital, NEVSOM)
Record Dates: First submitted 2023-04-14; First posted 2023-05-25 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Attention Deficit Hyperactivity Disorder; Executive Dysfunction
Keywords: adolescents; Goal Management Training
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Goal management training (Experimental): Cognitive rehabilitation:14 hours of GMT in groups of 4-6 participants, administered following a script with accompanying PowerPoint slides and participant workbooks, over the course of 7 weeks (one 2-hour session per week). In addition, the participants receive Treatment as Usual
  Interventions: Behavioral: Goal Management training
- Treatment as Usual (No Intervention): Norway has established clinical guidelines for ADHD assessment and treatment in public health, emphasizing psychoeducation, parent management training, school counseling, and pharmacological treatment adapted to the needs of each patient

INTERVENTIONS:
Behavioral: Goal Management training — metacognitive group intervention
  Arms: Goal management training

SUMMARY:
The goal of this clinical trial is to evaluate an evidence-based, non-pharmacological treatment alternative: Goal Management Training (GMT) for adolescents with Attention-Deficit/Hyperactivity Disorder (ADHD). The main questions we aim to answer are:

1. Is GMT more effective than Treatment as Usual (TAU) in improving executive functioning in adolescents with ADHD?
2. Is GMT more effective than TAU in improving emotional health and social functioning in adolescents with ADHD?
3. Which clinical or cognitive characteristics are associated with treatment response?
4. Do medication, age, gender, and functional status at intake influence treatment response and long-term outcomes?
5. Are genetic (e.g. polygenic risk scores) and brain imaging data (e.g. estimates of brain maturation based on structural MRI or resting-state functional magnetic resonance imaging (fMRI) brain connectivity) relevant clinical predictors for treatment response and long-term outcomes?

DETAILED DESCRIPTION:
ADHD is characterized by impaired executive functions (EFs). EFs are brain functions that allow us to direct our attention, retain relevant information, and ignore distractions in order to achieve our daily goals. Impairments in EF are associated with poorer academic achievement and vocational functioning, psychopathology symptoms, emotional and social problems, as well as lower quality of life in children and adolescents with ADHD. Furthermore, pharmacological treatment has not been shown to significantly improve EF difficulties, and there is still a considerable knowledge gap regarding the efficacy of non-pharmacological treatment for ADHD. Additionally, the research is often limited by short follow-up periods and few outcome measures.

We propose a randomized controlled trial, comparing a seven-week non-pharmacological cognitive remediation program designed to improve EFs; Goal Management Training (GMT), to treatment-as-usual (TAU) for 120 adolescents with ADHD. The primary outcome is executive function behaviors in the school and home environments (Behavior Rating Inventory of Executive Function 2, parent report). Secondary outcomes include neuropsychological tests, mental health, quality of life, and social deficit symptoms. Participants will be assessed at baseline, after 12 weeks, and 12- and 24 months post-treatment. In addition, we will collect biological samples and brain MRI data in a sub-sample, which will allow us to test whether genetic (e.g. polygenic scores) and brain imaging data collected at baseline (e.g. estimates of brain maturation based on structural MRI or resting-state fMRI brain connectivity) are relevant clinical predictors for treatment response and long-term outcomes. If sample size allows, these analyses will be purely exploratory, and the relevant measures will not be specified in this registration.

The expected main benefit of the described study is to provide evidence-based non-pharmacological treatment to a vulnerable group, potentially improving life-long function and adherence to education, work, and social life.

During the autumn of 2024, a qualitative interview will be conducted with a few participants who have completed GMT, and the co-therapists will participate in a focus group interview. The purpose is to complement the quantitative data from the main study with qualitative data on how GMT is experienced by participants and therapists. This sub-study has been approved by the ethics committee and data protection authorities.

ELIGIBILITY:
Inclusion Criteria:

1. Adolescents with a diagnosis of ADHD (ICD-10, DSM-5).
2. Aged 12-18 years. We will include irrespective of concurrent or previous pharmacological treatment.

Exclusion Criteria:

1. Severe depression, suicidality, psychosis, bipolar disorder without stable medication and current substance abuse
2. Organic brain injury or verified neurological disease (3) cognitive or medical impairments that have affected or are affecting the capacity to attend regular school.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Parent-Reported Behavior Rating Inventory of Executive Function - Second Edition (BRIEF-2). | Change from Baseline up to 24 months (Assessed at Baseline, after 12 weeks, after 12 months, and after 24 months).
  Rating inventory assessing executive function in daily life. Higher scores indicate greater executive dysfunction. The total score ranges from 86 - 258.

SECONDARY OUTCOMES:
Change in Self-Reported Behavior Rating Inventory of Executive Function - Second Edition (BRIEF-2). | Change from Baseline up to 24 months (Assessed at Baseline, after 12 weeks, after 12 months, and after 24 months).
  Rating inventory assessing executive function in daily life. Higher scores indicate greater executive dysfunction. The total score ranges from 80 - 240.
Change in Teacher-Reported Behavior Rating Inventory of Executive Function - Second Edition (BRIEF-2). | Change from Baseline up to 12 weeks (Assessed at Baseline, and after 12 weeks).
  Rating inventory assessing executive function in daily life. Higher scores indicate greater executive dysfunction. The total score ranges from 86 - 258.
Change in Attention Span task from Cognitive Assessment at Bedside for IPad (CABPad). | Change from Baseline up to 12 weeks (Assessed at Baseline, and after 12 weeks).
  Performance-based Executive functioning tests: To assess simple attention span. The scoring is based on the number of objects remembered. More objects indicate higher attention span.
Change in Working Memory task from Cognitive Assessment at Bedside for IPad (CABPad). | Change from Baseline up to 12 weeks (Assessed at Baseline, and after 12 weeks).
  Performance-based Executive functioning test: To assess working memory. The scoring is based on the number of objects remembered. More objects indicate a better working memory.
Change in Arrow Stroop task from Cognitive Assessment at Bedside for IPad (CABPad). | Change from Baseline up to 12 weeks (Assessed at Baseline, and after 12 weeks).
  Performance-based Executive functioning test: To investigate executive control of attention, more specifically cognitive impulse control. Scoring is based on reaction time and the number of incorrect/correct responses.
Change in Symbol Digit Coding (Mental and Visuo-Motor Speed) task from Cognitive Assessment at Bedside for IPad (CABPad). | Change from Baseline up to 12 weeks (Assessed at Baseline, and after 12 weeks).
  Performance-based Executive functioning test: To investigate mental and visuo-motor speed. Scoring is based on reaction time and the number of incorrect/correct responses.
Change in Parent-Reported Achenbach System of Empirically Based Assessment (ASEBA). | Change from Baseline up to 24 months (Assessed at Baseline, after 12 weeks, and after 24 months).
  Assessment rating adaptive and maladaptive functioning. Higher scores indicate greater difficulty. The total score ranges from 0 - 224.
Change in Self-Reported Achenbach System of Empirically Based Assessment (ASEBA). | Change from Baseline up to 24 months (Assessed at Baseline, after 12 weeks, and after 24 months).
  Assessment rating adaptive and maladaptive functioning. Higher scores indicate greater difficulty. The total score ranges from 0 - 224.
Change in Parent-Reported Weiss Functional Impairment Rating Scale (WFIRS-P). | Change from Baseline up to 24 months (Assessed at Baseline, after 12 weeks, and after 24 months).
  Rating inventory that evaluates the extent to which an individual's ability to function is impaired. The 50-item scale uses a Likert scale, such that any item rating 2 or 3 is clinically impaired. The total score ranges from 0 - 150.
Change in Parent-Reported ADHD Rating scale (ADHD-RS-IV Home). | Change from Baseline up to 24 months (Assessed at Baseline, after 12 weeks, and after 24 months).
  Rating inventory that detects ADHD symptoms in children and adolescents reported by parents. The 18-item scale generates a total score between 0 - 54, where the higher score indicates greater difficulty.
Change in Teacher-Reported ADHD Rating scale (ADHD-RS-IV School). | Change from Baseline up to 12 weeks (Assessed at Baseline, and after 12 weeks).
  Rating inventory that detects ADHD symptoms in children and adolescents. The 18-item scale generates a total score between 0 - 54, where the higher score indicates greater difficulty.
Change in Parent-Rated Pediatric Quality of Life Inventory (PedsQL). | Change from Baseline up to 24 months (Assessed at Baseline, after 12 weeks, and after 24 months).
  Measurement of health-related quality of life. The 23-item scale generates a total score between 0-100, where 100 points indicate optimal quality of life.
Change in Self-Rated Pediatric Quality of Life Inventory (PedsQL). | Change from Baseline up to 24 months (Assessed at Baseline, after 12 weeks, and after 24 months).
  Measurement of health-related quality of life.The 23-items scale generates a total score between 0-100, where 100 points indicate optimal quality of life.
Change in Goal Attainment Scaling (GAS). | Change from Baseline up to 12 weeks (Assessed at Baseline, and after 12 weeks).
  Method of rating performance based on a criterion-referenced scale with defined anchor points. If the patient achieves the expected level, this is scored at 0. If they achieve a better than expected outcome this is scored at: +1 (somewhat better), +2 (much better). If they achieve a worse than expected outcome this is scored at: -1 (somewhat worse), or -2 (much worse). The patient and the clinician decide this score together.
Change in Children's Global Assessment Scale (CGAS). | Change from Baseline up to 12 weeks (Assessed at Baseline, and after 12 weeks).
  Measure of a child's or adolescent's psychosocial functioning on a scale from 1 (lowest functioning) to 100 (superior functioning in all areas). Rated by an independent observer.

CONTACTS AND LOCATIONS:
Overall Officials: Merete G Øie, PhD, Principal Investigator — Department of Psychology, Faculty of Social Sciences, University of Oslo
Locations (2):
- Norway (2):
  - Innlandet hospital trust, Brumunddal, Brumunddal
  - Lovisenberg Diakonale Hospital, Oslo, Oslo County

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol